## Fu Jen Catholic University Institutional Review Board

510 Chung Cheng Rd, Hsinchuang District, New Taipei City 242062, Taiwan TEL: 886-2-2905-6277,FAX: 886-2-2903-3546

TEL: 886-2-2905-62/7,FAX: 886-2-2905-554

## Certificate of Approval

I. FJU-IRB NO: C112161

- II. Study Institution(s): Department of Exercise and Health Science/ National Taipei University of Nursing and Health Sciences
- III. Investigator: Professor Wen Ching Huang

IV. Research team member(s):

1. Fan, Ching-Wen/Department of Exercise and Health Science/National Taipei University of Nursing and Health Sciences

2. Huang, Siao-Fen/Department of Exercise and Health Science/National Taipei University of Nursing and Health Sciences

V. Title of protocol: The effects of interactive stampede exercise training on elderly physical activities, life quality, and physical fitness

VI. Protocol Version:第3版,2024/06/03

- VII. Informed Consent Form: 第5版, 2024/06/13
- VIII. Place of execution(s): National Taipei University of Nursing and Health Sciences
- IX. Study Tools:

Questionnaire(s):

- 1. 身體活動準備度問卷/第2版,2024/05/21
- 2. IPAQ台灣活動量調查/第1版,2024/04/25
- 3. 生活品質量表-台灣版/第1版, 2024/04/25

Recruitment Version:招募廣告/第3版,2024/06/03

- X. Frequency of Interim Report: One Year
- XI. Study Approval Period: 2024/06/13~2025/06/12

in chen

The protocol has been approved by the Institutional Review Board of Fu Jen Catholic University. The committee is organized under, and operates in accordance with Regulations of Fu Jen Catholic University and governmental laws and regulations. Continuing Review Application should be submitted to Institutional Review Board no later than 4 weeks before current approval expired. The investigator is required to report protocol amendment and serious adverse events in accordance with the Fu Jen Catholic University and governmental laws and regulations.

Chair's Signature

Institutional Review Board

06 114 12024

Date (mm / dd / yyyy)